CLINICAL TRIAL: NCT02057354
Title: Aerobic Exercise, Neurotrophins, and fMRI of Hippocampal Function and Structure
Brief Title: Neuroimaging Study of Exercise and Memory Function
Acronym: EMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Karin Schon, Assisstant Professor, Department of Anatomy & Neurobiology, BUSM, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-32635; R00AG036845 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Aging
Keywords: Brain; Brain-Derived Neurotrophic Factor; Brain Mapping; Cognition; Exercise; Hippocampus; Hydrocortisone; Learning; Memory; Magnetic Resonance Imaging; Nerve Growth Factors; Neuroimaging; Physical Endurance; Physical Fitness; Resistance Training; Walking
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Sedentary Young Adults (Active Comparator): Participants 18-35 years of age will be randomized to either aerobic or non-aerobic exercise training.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Non-Aerobic Exercise
- Healthy Sedentary Older Adults (Experimental): Participants 55-85 years of age will be randomized to either aerobic or non-aerobic exercise training.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Non-Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — The goal of the aerobic exercise training is to increase aerobic endurance. Walking on treadmill at moderate intensity with grade adjusted. Exercise tailored to individual ability level.
  Other Names: Endurance Training
Behavioral: Non-Aerobic Exercise — The goal of this training is to improve overall muscle strength, balance and flexibility. Participants will do strength, balance and stretching exercises. Exercises tailored to individual ability level.
  Other Names: Strength, balance, stretching

SUMMARY:
The investigators are examining the effects of exercise and cardiovascular fitness on cognitive processes, brain function, and the amount of several proteins in the blood. These proteins include a hormone called cortisol, also known as the "stress hormone," and a growth factor called "brain-derived neurotrophic factor" (BDNF). The "stress hormone" cortisol is produced by the adrenal glands. Stress, exercise, obesity, and other factors may influence cortisol levels. BDNF is a protein that promotes the health of nerve cells in the brain and in the body. It plays a role in the growth, maturation, and maintenance of these cells. The amount of this protein in blood samples is therefore an indicator of healthy nerve cell function. Here, the investigators are investigating if exercise improves brain function by changing BDNF levels. Participation in this research study will take approximately 4 months. During this time, participants will make four initial study visits. The first visit is for informed consent and screening, the second and third visits are for baseline fitness testing, and the fourth visit is for a blood draw, cognitive testing, and a functional Magnetic Resonance Imaging (fMRI) exam. Functional MRI is a brain imaging technique that uses a magnetic field to "take pictures" of the brain while a person performs a given task. It will take up to approximately three weeks to complete these initial four study visits. Following the four initial study visits, the exercise-training program will begin. Participants will be randomized to one of two training programs: an aerobic exercise program and a non-aerobic exercise program consisting of strengthening, balance and stretching exercises. The exercise training program will last 12 weeks. There will be three one-hour exercise sessions per week. After completion of the exercise-training program, participants will attend three follow-up study visits. The first two follow-up visits are for fitness testing. The third and final follow-up visit is for a blood draw, cognitive testing, and an MRI exam.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Age between 18-35 years or between 55-85 years
* Sedentary status (physically inactive)
* Generally healthy
* Native-English speaker

Exclusion Criteria:

* Diagnosis of severe anemia
* Past or present condition that affect cognitive functioning:

  1. learning disability
  2. neurological disorders or conditions (movement disorder, history of head trauma or stroke, epilepsy, etc.)
  3. psychiatric disorders or conditions (depression, anxiety disorder, etc.)
* Poor vision that cannot be corrected with glasses or contact lenses
* Presence of an infection
* Diagnosis of kidney failure
* Diagnosis of liver disease
* Diagnosis of thyrotoxicosis/hyperthyroidism
* Diagnosis of cancer
* Past or present conditions that are counter indicators for participation in cardio-respiratory fitness assessment and physical exercise:

  1. heart (e.g. heart attack, arrhythmias, etc.)
  2. circulatory (e.g. uncontrolled hypertension, high cholesterol, etc.)
  3. respiratory conditions (e.g., asthma or lung conditions, such as chronic obstructive pulmonary disease, acute bronchitis, acute common cold, lung cancer, pneumonia, etc.)
  4. current musculoskeletal impairments (e.g. leg claudication, fractures, hemiplegia, chronic joint pain, arthritis, osteoporosis, not able to walk comfortably without assistance, etc.)
  5. diagnosis of electrolyte disorder or abnormality
  6. presence of diabetes mellitus
* Claustrophobia (fear of small, encloses spaces)
* Female subjects: breast-feeding or potentially pregnant
* Obesity
* Eating disorder
* Compulsive exercising
* Ferro-magnetic metal in or on the body that cannot be removed (e.g. pacemaker, defibrillator, permanent tattoo or eyeliner with metallic specks)
* Prescription medication or other drugs that are cardio-active
* Prescription medication or other drugs that are psycho-active
* Drug abuse or alcohol misuse
* Regularly exercising
* Unavailable for the approximately 4-month duration of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
MRI | 1.5 to 2 hours each at Visits 4 and 43
  Measurement of brain activity during task performance and measurement of change in regional brain volumes.
Serum BDNF level | 5 minutes each at Visits 4 and 43
  Fasting blood draw on same day of MRI to measure change in serum BDNF from baseline to follow-up
Memory test performance | 1.5 to 2 hours each at Visits 4 and 43
  Participants will perform recognition memory tests during and after functional MRI. Measurements include baseline-to-follow-up change in reaction times and accuracy.

SECONDARY OUTCOMES:
Aerobic capacity and muscle strength | 80 min each at Visits 2, 3, 41 and 42
  Participants will perform two treadmill tests and several muscle strength tests to estimate baseline-to-follow-up change in aerobic capacity, measure change in time on treadmill, and determine change in muscle strength.

OTHER OUTCOMES:
Blood cortisol levels | 5 min each at Visits 4 and 43
  Cortisol levels will be obtained from the blood sample drawn during baseline and follow-up.
Anthropometric measurements | 10 minutes each during Visits 2 and 41
  Anthropometric measurements include height, weight, and body mass index. Percent body fat will also be estimated.
Blood serum levels of other neurotrophins | 5 min each at Visit 4 and 43
  The blood draw will be used for other neurotrophins related to exercise and cognition.
Neuropsychological test performance | 15-30 minutes each at Visits 4 and 43
  Baseline-to-follow-up change in performance of the Wechsler Adult Intelligence Scale-IV subtests

CONTACTS AND LOCATIONS:
Overall Officials: Karin Schon, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kern KL, Storer TW, Schon K. Cardiorespiratory fitness, hippocampal subfield volumes, and mnemonic discrimination task performance in aging. Hum Brain Mapp. 2021 Mar;42(4):871-892. doi: 10.1002/hbm.25259. Epub 2020 Dec 16. PMID 33325614
- [Derived] Nauer RK, Dunne MF, Stern CE, Storer TW, Schon K. Improving fitness increases dentate gyrus/CA3 volume in the hippocampal head and enhances memory in young adults. Hippocampus. 2020 May;30(5):488-504. doi: 10.1002/hipo.23166. Epub 2019 Oct 7. PMID 31588607